CLINICAL TRIAL: NCT03846466
Title: A Phase 1 Randomized, Double-Blind, Placebo-Controlled, Single Dose or Multiple Dose Study of KHK4323 in Healthy Volunteers, and Subjects With Atopic Dermatitis
Brief Title: Study of KHK 4323 in Healthy Volunteers and Subjects With Atopic Dermatitis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study terminated for safety reasons.
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4323-001
Record Dates: First submitted 2019-02-17; First posted 2019-02-19 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (18):
- Part1 Dose 1A (Experimental): Single administration
  Interventions: Drug: KHK4323 IV/S
- Part1 Dose 1P (Placebo Comparator): Single administration
  Interventions: Drug: Placebo IV/S
- Part1 Dose 2A (Experimental): Single administration
  Interventions: Drug: KHK4323 IV/S
- Part1 Dose 2P (Placebo Comparator): Single administration
  Interventions: Drug: Placebo IV/S
- Part1 Dose 3A (Experimental): Single administration
  Interventions: Drug: KHK4323 IV/S
- Part1 Dose 3P (Placebo Comparator): Single administration
  Interventions: Drug: Placebo IV/S
- Part1 Dose 4A (Experimental): Single administration
  Interventions: Drug: KHK4323 IV/S
- Part1 Dose 4P (Placebo Comparator): Single administration
  Interventions: Drug: Placebo IV/S
- Part1 Dose 5A (Experimental): Single administration
  Interventions: Drug: KHK4323 SC/S
- Part1 Dose 5P (Placebo Comparator): Single administration
  Interventions: Drug: Placebo SC/S
- Part1 Dose 6A (Experimental): Single administration
  Interventions: Drug: KHK4323 IV/S
- Part1 Dose 6P (Placebo Comparator): Single administration
  Interventions: Drug: Placebo IV/S
- Part1 Dose 7A (Experimental): Single administration
  Interventions: Drug: KHK4323 IV/S
- Part1 Dose 7P (Placebo Comparator): Single administration
  Interventions: Drug: Placebo IV/S
- Part2 Dose 1A (Experimental): Multiple administration
  Interventions: Drug: KHK4323 IV/M
- Part2 Dose 1P (Placebo Comparator): Multiple administration
  Interventions: Drug: Placebo IV/M
- Part2 Dose 2A (Experimental): Multiple administration
  Interventions: Drug: KHK4323 IV/M
- Part2 Dose 2P (Placebo Comparator): Multiple administration
  Interventions: Drug: Placebo IV/M

INTERVENTIONS:
Drug: KHK4323 IV/S — IV / Single administration
  Arms: Part1 Dose 1A; Part1 Dose 2A; Part1 Dose 3A; Part1 Dose 4A; Part1 Dose 6A; Part1 Dose 7A
Drug: KHK4323 SC/S — SC / Single administration
  Arms: Part1 Dose 5A
Drug: KHK4323 IV/M — IV / Multiple administration
  Arms: Part2 Dose 1A; Part2 Dose 2A
Drug: Placebo IV/S — IV / Single administration
  Arms: Part1 Dose 1P; Part1 Dose 2P; Part1 Dose 3P; Part1 Dose 4P; Part1 Dose 6P; Part1 Dose 7P
Drug: Placebo IV/M — IV / Multiple administration
  Arms: Part2 Dose 1P; Part2 Dose 2P
Drug: Placebo SC/S — SC / Single administration
  Arms: Part1 Dose 5P

SUMMARY:
Part 1: To investigate the safety and tolerability of intravenous (IV) or subcutaneous (SC) administration of a single dose of KHK4323 to Japanese or Caucasian healthy adult males in a double-blind, placebo-controlled study.

Part 2: To investigate the safety and tolerability of intravenous (IV) administration of repeated doses of KHK4323 to atopic dermatitis patients in a double-blind, placebo-controlled study.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

* Japanese or Caucasian male aged 20 to under 45 years old at the time consent was obtained
* BMI ≥ 18.5 to < 30.0 at time of screening tests

Part 2:

* Men and women aged 18 years or older at the time of consent
* Patients with EASI ≥ 16 in pre-administration testing
* Patients with IGA of "3: Moderate" or higher in pre-administration testing
* Patients with BSA ≥ 10% at screening in pre-administration testing

"Exclusion Criteria:

Part 1:

* Persons with existing respiratory disease, heart disease, gastrointestinal disease, kidney disease, or liver disease
* Persons confirmed to have a bacterial, viral, fungal, or parasitic infection within 28 days prior to obtainment of consent
* Persons who have contracted an infectious disease requiring hospitalization or IV administration of an antibiotic within 6 months prior to obtainment of consent
* Persons who have been treated with a biological preparation (antibody, etc.) or have been administered an investigational drug within 6 months prior to the obtainment of consent
* Persons who have used a medication (including over-the-counter drugs, topical agents, vitamins, and herbal medicines) within 2 weeks prior to obtainment of consent (for an immunosuppressant drug, within 60 days)
* Persons who routinely smoke an average of more than 10 cigarettes a day (to be confirmed in interview at time of screening tests) or cannot follow the rules regarding smoking during the clinical trial period

Part 2:

* Patients with severe complications judged to affect the implementation and evaluation of the study in the opinion of the investigator or sub-investigator. Includes but is not limited to the following. Severe cardiovascular disease (e.g., class III or IV according to New York Heart Association functional classification), poorly controlled diabetes mellitus (HbA1c > 8.5%), poorly controlled hypertension, liver disease with severity of moderate or higher (e.g., class B or C according to Child-Pugh classification), kidney disease, respiratory disease, gastrointestinal disease, blood dyscrasia, central nervous system disease, psychiatric disease, autoimmune disease, etc.
* Patients observed to have one of the following laboratory test abnormalities in screening tests

  * Neutrophil count: < 1500/μL
  * Serum creatinine: > 1.5 mg/dL
  * AST or ALT: > 2.5-fold the upper limit of the reference range
  * Other laboratory test abnormalities that the investigator or sub-investigator thinks could affect the completion or evaluation of the clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Part 1: from Day 1 through at most Day 169, Part 2: from Day 1 through at most Day 225
  For adverse events that occurred after administration of the investigational drug, number of subjects with AEs and occurrence frequency are classified by MedDRA PT and SOC and shown according to dose group.

SECONDARY OUTCOMES:
Profile of pharmacokinetics of serum KHK4323 concentration in Part 1 | Day 1 (pre-dose, 1, 6 hours after the start of administration) Day 2, Day 3, Day 4, Day 8, Day 15, Day 29, Day 43, Day 57, Day 71, Day 85, Day 99, Day 113, Day 127, Day 141, Day 169
  Anti-KHK4323 antibodies
Profile of pharmacokinetics of serum KHK4323 concentration in Part 2 | Day 1( pre-dose, 1 hours after the start of administration), Day 8, Day 15, Day 29,Day 43, Day 57, Day 85, Day 113, Day 169, Day 225
  Anti-KHK4323 antibodies

OTHER OUTCOMES:
Change from baseline in Eczema Area and Severity Index (EASI) | Part2: Day1(Pre-dose), Day 15, Day 29,Day 43, Day 57, Day 85, Day 113, Day 141, Day 169, Day 197, Day 225
Percent change in Eczema Area and Severity Index (EASI) | Part2: Day1(Pre-dose), Day 15, Day 29,Day 43, Day 57, Day 85, Day 113, Day 141, Day 169, Day 197, Day 225
Change from baseline in Body surface area (BSA) of involvement of Atopic dermatitis | Part2 Day1(Pre-dose), Day 15, Day 29, Day 43, Day 57, Day 85, Day 113, Day 141, Day 169, Day 197, Day 225
Percent change in Body surface area (BSA) of involvement of Atopic dermatitis | Part2 Day1(Pre-dose), Day 15, Day 29, Day 43, Day 57, Day 85, Day 113, Day 141, Day 169, Day 197, Day 225
The number of subjects with IGA of 0 or 1 and improvement of 2 points or more over baseline score (IGA responders) | Part2 Day1(Pre-dose), Day 15, Day 29, Day 43, Day 57, Day 85, Day 113, Day 141, Day 169, Day 197, Day 225
The percentage of subjects with IGA of 0 or 1 and improvement of 2 points or more over baseline score (IGA responders) | Part2 Day1(Pre-dose), Day 15, Day 29, Day 43, Day 57, Day 85, Day 113, Day 141, Day 169, Day 197, Day 225

CONTACTS AND LOCATIONS:
Locations (1):
- Osaka Pharmacology Clinical research Hospital, Osaka, Japan